CLINICAL TRIAL: NCT03486301
Title: Phase 1 Open-Label Dose Escalation Study of BDB001 as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: BDB001-101: Clinical Study of BDB001 as a Mono-therapy or in Combination With Pembrolizumab
Acronym: EIK1001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BDB001-101; KEYNOTE-914 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2018-02-28; First posted 2018-04-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid
Keywords: TLR7/8; Immuno-oncology; EIK1001
MeSH Terms: conditions — Neoplasms | interventions — BDB001; pembrolizumab

STUDY DESIGN:
Intervention Model Description: BDB001 followed by combination treatment with KEYTRUDA®
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Agent BDB001 (EIK1001) (Experimental): A single subject will be enrolled at each dose level in the single agent arm until any ≥ Grade 2 treatment-emergent adverse event (TEAE) is observed in the first cycle.
  Then dosage escalation will follow a traditional 3+3 dose escalation design.
  Each successive group of patients will be enrolled at an incrementally higher dosage until the Maximum Tolerable Dose (MTD) or Recommended Phase 2 Dose (RP2D) of single agent BDB001 is reached.
  Interventions: Drug: BDB001 (EIK1001)
- BDB001 in Combination with Pembrolizumab (Experimental): In the combination arm of the study, a standard 3+3 dose escalation design will be utilized for all dose levels.
  When the MTD or RP2D of single agent BDB001 is reached, the first dose level cohort of the combination arm will begin. Once the MTD or RP2D in combination has been determined, twenty additional subjects will be enrolled in the expansion phase of the study.
  Interventions: Drug: BDB001 (EIK1001); Drug: Pembrolizumab

INTERVENTIONS:
Drug: BDB001 (EIK1001) — BDB001 (EIK1001) is an immunotherapy agent.
Drug: Pembrolizumab — Pembrolizumab is a potent humanized monoclonal antibody with high specificity of binding to the PD 1 receptor. Pembrolizumab has an acceptable preclinical safety profile and is approved as an IV therapy for a variety of advanced malignancies.
  Arms: BDB001 in Combination with Pembrolizumab

SUMMARY:
Phase 1 Open-Label Dose Escalation Study of BDB001 as a Single Agent and in combination with Pembrolizumab in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This clinical trial is a study of an experimental drug called BDB001. BDB001 is a Toll-like receptor (TLR) agonist that activates the immune system.

The primary objectives of this study are to evaluate the safety and tolerability of BDB001 as a single agent and in combination with pembrolizumab and to determine the maximum tolerated dose (MTD) or the recommended Phase 2 dose (RP2D) when given in combination with pembrolizumab in subjects with advanced solid tumors.

This is a multi-center, open-label, dose escalation/dose expansion Phase 1 study of BDB001 as a single agent and in combination with pembrolizumab in subjects with histologically-confirmed, incurable, unresectable or metastatic solid tumors that have relapsed or are refractory to standard therapies or for whom there is no approved therapy.

The study will be conducted in two separate but independent dose escalation arms: a single agent arm (BDB001 alone) and a combination arm (BDB001 in combination with pembrolizumab).

Participants will be allowed to continue treatment beyond study termination until occurrence of significant treatment-related toxicity, progressive disease or discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Be 18 years of age on day of signing informed consent
2. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors who have disease progression after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment. Note: there is no limit to the number of prior treatment regimens
3. A male participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
4. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP)
   2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment • A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year, when used consistently and correctly)
5. Evidence of progressive disease (PD) within 3 months of signing the informed consent form
6. Have measurable disease per irRECIST as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
7. Eastern Cooperative Oncology Group (ECOG) score of 0 - 2
8. Minimum life expectancy of 3 months
9. Have adequate organ function as defined by the protocol. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. A woman of child bearing potential who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
2. Prior exposure to TLR 7 agonists (e.g., GS-9620, imiquimod, TMX 101, resiquimod, MEDI9197, 825A) and TLR 9 agonists (e.g., SD-101, IMO2125, MGN1703, GNKG168, DUK-CPG-001 and CMP-001) for treatment of the solid tumor the patient is currently being evaluated for treatment with BDB001.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher irAE
4. Received previous therapy for malignancy within 21 days prior to administration of study drug, including any investigational agents (other than BDB001), chemotherapy, immunotherapy, biological or hormonal therapy (6 weeks for nitrosoureas or mitomycin C)
5. Major surgery within 4 weeks of first dose of study drug
6. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
7. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
8. Currently receiving medications known to be strong inhibitors of CYP1A and CYP3A and strong/moderate inducers of CYP1A and CYP3A
9. Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
10. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 21 days prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
11. History within last 6 months of New York Heart Association Class III or IV heart failure, acute myocardial infarction, angina pectoris, uncontrolled arrhythmia, acute coronary syndromes, stent placement, uncontrolled hypertension
12. QTc interval value > 470 msec (using Fridericia's Correction)
13. Left ventricular ejection fraction (LVEF) < 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
14. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment (Kim 2017).
15. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
16. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
17. Known active hepatitis A, B or C. Subjects who are HBsAg+ and have DNA load < 2000 IU/mL (104 copies/mL) are eligible to participate in the study provided they meet the ALT and bilirubin inclusion criteria.
18. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
19. Has an active infection requiring systemic therapy
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
21. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
22. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
23. Has had an allogenic tissue/solid organ transplant
24. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
25. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
26. History of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: incidence of adverse events and any dose limiting toxicity | Up to 30 months
  Safety and tolerability of BDB001 as a single agent and in combination with pembrolizumab as measured by the incidence of adverse events and any dose limiting toxicity

SECONDARY OUTCOMES:
Determine Maximum Tolerated Dose | From first dose to 21 days after first dose for each patient (cycle 1)
  Determination of the maximum tolerated dose by assessing the frequency of BDB001-related and BDB001 and pembrolizumab-related adverse events using CTCAE version 4.03 to categorize adverse event severity
Radiographic Determination of Tumor Response after BDB001 Dosing | Every 63 days (3 cycles) up to 30 months after the first dose for each patient (each cycle is 21 days)
  Radiographic determination of tumor response in subjects dosed with BDB001 and BDB001 and pembrolizumab using irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Harry Raftopoulos, MD, Study Chair — Eikon Therapeutics
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Sarasota, Florida
  - Atlantic Health, Morristown, New Jersey
  - Tennessee Oncology, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No